CLINICAL TRIAL: NCT03128281
Title: A Single Center, Prospective, Randomized, Controlled Study to Evaluate Shoulder Pain, Cardiovascular Changes, Pulmonary Pressures and Perioperative Outcomes Related to the Use of the AirSeal® Insufflation System (AIS) at Low and Higher Pressure Pneumoperitoneum vs. Conventional Insufflation
Brief Title: Pneumoperitoneum Management With Low vs. Higher Pressure
Status: Withdrawn | Phase: Phase 2 | Type: Interventional
Why Stopped: Sponsor issue
Sponsor: M.D. Anderson Cancer Center (Other)
Collaborators: CONMED Corporation (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 2015-0973; NCI-2018-01330 (Registry Identifier: NCI CTRP)
Record Dates: First submitted 2017-04-20; First posted 2017-04-25 (Actual); Last update posted 2019-05-30 (Actual); Status verified 2019-05

CONDITIONS: Malignant Neoplasms of Female Genital Organs
Keywords: Malignant Neoplasms of Female Genital Organs; Laparoscopic gynecologic surgery; Robotic gynecologic surgery; AirSeal® Insufflation System; AIS; Conventional Insufflation System; CIS; Questionnaires; Surveys
MeSH Terms: interventions — Surveys and Questionnaires

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

ARMS (3):
- Conventional Insufflation System (CIS) (Experimental): Questionnaires completed 30 days before surgery, two (2) hours after surgery, when leaving the post-anesthesia care unit (PACU), and at hospital discharge.
  Conventional Insufflation System (CIS) used for pneumoperitoneum during laparoscopic/robotic surgery.
  Interventions: Behavioral: Questionnaires; Device: Conventional Insufflation System (CIS)
- ConMed AirSeal Insufflation System (AIS) at Low Pressure (Experimental): Questionnaires completed 30 days before surgery, two (2) hours after surgery, when leaving the post-anesthesia care unit (PACU), and at hospital discharge.
  ConMed AirSeal Insufflation System (AIS) at Low Pressure used for pneumoperitoneum during laparoscopic/robotic surgery.
  Interventions: Behavioral: Questionnaires; Device: ConMed AirSeal Insufflation System (AIS) at Low Pressure
- ConMed AirSeal Insufflation System (AIS) at Higher Pressure (Active Comparator): Questionnaires completed 30 days before surgery, two (2) hours after surgery, when leaving the post-anesthesia care unit (PACU), and at hospital discharge.
  ConMed AirSeal Insufflation System (AIS) at Higher Pressure used for pneumoperitoneum during laparoscopic/robotic surgery.
  Interventions: Behavioral: Questionnaires; Device: ConMed AirSeal Insufflation System (AIS) at Higher Pressure

INTERVENTIONS:
Behavioral: Questionnaires — Questionnaires completed 30 days before surgery, two (2) hours after surgery, when leaving the post-anesthesia care unit (PACU), and at hospital discharge.
  Questionnaires ask about pain level and any drugs taken for it. It should take about 5 minutes to complete.
  Other Names: Surveys
Device: Conventional Insufflation System (CIS) — CIS with pressure target of 15±1 mmHg used for pneumoperitoneum during laparoscopic/robotic surgery.
  Other Names: CIS
  Arms: Conventional Insufflation System (CIS)
Device: ConMed AirSeal Insufflation System (AIS) at Low Pressure — AIS with an insufflation pressure target of 9±1 mmHg used for pneumoperitoneum during laparoscopic/robotic surgery.
  Other Names: AIS
  Arms: ConMed AirSeal Insufflation System (AIS) at Low Pressure
Device: ConMed AirSeal Insufflation System (AIS) at Higher Pressure — AIS with an insufflation pressure target of 15±1 mmHg used for pneumoperitoneum during laparoscopic/robotic surgery.
  Other Names: AIS
  Arms: ConMed AirSeal Insufflation System (AIS) at Higher Pressure

SUMMARY:
The goal of this clinical research study is to compare the level of pain 2 hours after surgery in patients after the use of the AirSeal® Insufflation System (AIS) at a high or low pressure setting or the standard insufflator (the conventional insufflation system, or CIS). "Insufflation" is the creation of a pressure barrier of air/gas within the abdomen that allows the surgeon more space to work in.

DETAILED DESCRIPTION:
Baseline Visit:

If participant agrees to take part in this study, within 30 days before surgery, participant will be asked to complete a questionnaire about participant's pain level and any drugs participant may be taking for it. It should take about 5 minutes to complete.

Study Groups:

Participant will be randomly assigned to 1 of 3 groups (as in a roll of dice). This is done because no one knows if one study group is better, the same, or worse than the other group. Participant has an equal chance of being placed in each group. Participant will not know which group participant is assigned to.

* If participant is in Group 1, participant will have the CIS used during surgery.
* If participant is in Group 2, participant will have the AIS used at a lower pressure during surgery.
* If participant is in Group 3, participant will have the AIS used at a higher pressure during surgery.

Surgery:

Participant will then have surgery. Participant will sign a separate consent for the surgery that explains the procedure, the risks of the surgery, and the risks of CIS.

Blood (about 3 teaspoons each time) will be collected 1 time before surgery, 2 times during surgery, and 1 time after surgery is completed. Routine tests and tests to learn how participant's body reacts to inflammation will be performed on this blood.

Questionnaires:

After surgery, participant will complete the questionnaire about participant's pain level and any drugs participant is taking. Participant will complete this questionnaire:

* Two (2) hours after surgery,
* When participant leaves the post-anesthesia care unit (PACU), and
* When participant is discharged from the hospital

If participant is discharged the same day as participant's surgery, participant will be called by the study staff to answer the questionnaire the following day.

Length of Study Participation:

Participation in the study will be over after participant completes the questionnaire after participant is discharged, unless participant agrees to complete additional optional questionnaires.

This is an investigational study. Both AirSeal® insufflation system (AIS) and conventional insufflation systems (CIS) are FDA approved and commercially available. It is investigational to compare the effects of high and low pressures using the AIS.

Up to 240 participants will be enrolled in this study. All will take part at MD Anderson.

ELIGIBILITY:
Inclusion Criteria:

1. All gynecologic laparoscopic/robotic surgeries EXCEPT diagnostic laparoscopies
2. 18-80 years of age
3. Capable and willing to provide Informed consent
4. Acceptable candidate for laparoscopic/robotic GYN surgery as per discretion of the surgeon
5. If patient agrees to participate in the optional patient reported outcomes portion of the study, patient must be English speaking and willing to complete the MD Anderson Symptom Inventory (MDASI) questionnaires

Exclusion Criteria:

1. Active cutaneous infection or inflammation
2. Pre-existing active or untreated immunodeficiency disorder and/or chronic use of systemic steroids
3. Uncontrolled diabetes mellitus
4. Severe co-existing morbidities having a life expectancy of less than 30 days
5. Significant anemia with hemoglobin level less than 7 g/dL or a hematocrit less than 21%
6. Females who are pregnant or lactating
7. Patients presenting with ascites
8. Patients with Chronic Pain Syndrome or requiring/using chronic pain medications
9. Patients undergoing diagnostic laparoscopy
10. Patients planning to undergo hand-assisted laparoscopy
11. Severe comorbidities (atrial fibrillation, pulmonary hypertension, etc...)

Ages: 18 Years to 80 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes
Enrollment: 0 (Actual)
Dates: Start 2018-07 (Estimated); Primary Completion 2021-07 (Estimated); Study Completion 2022-07 (Estimated)

PRIMARY OUTCOMES:
Incidence of Shoulder Pain After Laparoscopic/Robotic Surgery | Post-operative day 1
  Incidence of shoulder pain defined by a positive (>0) score for an 11-point pain intensity numeric rating scale (PI-NRS).

CONTACTS AND LOCATIONS:
Overall Officials: Pedro T. Ramirez, MD, Principal Investigator — M.D. Anderson Cancer Center

REFERENCES:
- See also: University of Texas MD Anderson Cancer Center Website — http://www.mdanderson.org